CLINICAL TRIAL: NCT01307553
Title: OVER AND UNDER/ANEUGRAFT PERICARDIUM COVERED STENT Long Term Follow Up Registry
Acronym: Sleeve III
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ITGI Medical (Industry)
Responsible Party: VP Medical Affairs, ITGI Medical
Other Study IDs: Sleeve III
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Diseased Saphenous Vein Grafts; Aneurysmal Coronary Arteries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PCS Group
  Interventions: Device: Pericardium Covered Stent

INTERVENTIONS:
Device: Pericardium Covered Stent — Percutaneous implantation of pericardium covered stent
  Other Names: Over and Under; Aneugraft

SUMMARY:
The purpose of this study is to track the clinical safety and effectiveness of the Pericardium Covered Stent in "real world" use.

DETAILED DESCRIPTION:
This is a multi-center registry of 75 patients treated with the Over and Under/Aneugraft Pericardium Covered Stent (PCS) (IGTI, Israel). The registry will involve the collection of demographic, clinical, and angiographic data on the treated patient population, including in-hospital, 30 day, 6-month, 1 year, 2 years and 3 years clinical follow-up data.

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 18 years
* Patient must be available for follow-up
* Patient must be fully informed, provided with the patient information sheet and sign the Informed Consent Form prior to the procedure.
* The lesion to be treated should be suitable for treatment with a PCS in that:

  * A. A suitable length and diameter PCS should be available
  * B. For SVG disease a single or multiple PCS may be used
  * C. For native coronary artery aneurysms the operator should be confident that the aneurysm may be excluded by the implantation of a single PCS

Exclusion Criteria:

* Significant co-morbidity precluding clinical follow-up.
* Pregnancy; pregnancy test negative in women with child bearing potential
* Acute ST-elevation myocardial infarction within the preceding 48 hours
* Previous stent implantation in the target vessel
* Left main coronary artery disease
* Contra-indication to dual anti-platelet therapy.
* Planned surgery which will lead to discontinuation of antiplatelet therapy
* Thrombocytopenia (<100,000/mm3)
* Ejection fraction <30%.
* Renal failure (creatinine >180 µmol/L [2 mg/dL])
* Prior brachytherapy
* Recipient of heart transplant
* Acute infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for PCI.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-10 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
MACE (Major Adverse Clinical Events) | 6 months

SECONDARY OUTCOMES:
MACE | 30 days, 1 Year, 2 Years, 3 Years
  MACE is a composite end point of cardiac death, myocardial infarction and target vessel revascularisation (TVR).
  Each one of the MACE components will be recorded separately
Hospital readmission due to cardiac reason. | 30 days, 6 months. 1 Year, 2 Years, 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Asif Qasim, Principal Investigator — King's College Hospital NHS Trust; Morris Mosseri, MD, Principal Investigator — Sapir Health Center, Cfar Saba, Israel
Locations (2):
- Sapir Health Center, Cfar Saba, Israel
- Kings College Hospital, London, United Kingdom

REFERENCES:
- [Background] Siregar S, Hoseyni Guyomi S, van Herwerden LA. Covered stents in giant coronary artery aneurysm. Eur Heart J. 2010 Nov;31(22):2823. doi: 10.1093/eurheartj/ehq267. Epub 2010 Jul 30. No abstract available. PMID 20675659
- [Background] Malkin C, Gunn J. A big cover-up. Heart. 2009 Aug;95(16):1354. doi: 10.1136/hrt.2009.171843. No abstract available. PMID 19638513
- [Background] Wykrzykowska JJ, Gutierrez-Chico JL, van Geuns RJ. "Over-and-under" pericardial covered stent with paclitaxel balloon in a saphenous vein graft. Catheter Cardiovasc Interv. 2010 May 1;75(6):964-6. doi: 10.1002/ccd.22412. PMID 20432403
- [Background] Tyczynski P, Kukreja N, van Geuns RJ, Wykrzykowska JJ, Sheppard MN, Di Mario C. Optical coherence tomography for the assessment of pericardium covered stents for the treatment of degenerated saphenous vein grafts. EuroIntervention. 2010 May;6(1):78-85. PMID 20542801
- [Background] Jokhi PP, McKenzie DB, O'Kane P. Use of a novel pericardial covered stent to seal an iatrogenic coronary perforation. J Invasive Cardiol. 2009 Oct;21(10):E187-90. PMID 19805849
- [Background] Hayat SA, Ghani S, More RS. Treatment of ruptured coronary aneurysm with a novel covered stent. Catheter Cardiovasc Interv. 2009 Aug 1;74(2):367-70. doi: 10.1002/ccd.21937. PMID 19642186
- [Background] Colombo A, Almagor Y, Gaspar J, Vonderwalde C. The pericardium covered stent (PCS). EuroIntervention. 2009 Aug;5(3):394-9. doi: 10.4244/v5i3a61. No abstract available. PMID 19736166
- [Background] Heper G, Barcin C, Iyisoy A, Tore HF. Treatment of an iatrogenic left internal mammary artery to pulmonary artery fistula with a bovine pericardium covered stent. Cardiovasc Intervent Radiol. 2006 Sep-Oct;29(5):879-82. doi: 10.1007/s00270-005-0149-2. PMID 16736101
- [Background] Gaspar J, Martinez-Rios MA, Vonderwalde C, Rosas M, Ban-Hayashi E, Eidt-Lidt G, Kuri J. Pericardium-covered stent for septal myocardial ablation in hypertrophic obstructive cardiomyopathy. Catheter Cardiovasc Interv. 1999 May;47(1):73-9. doi: 10.1002/(SICI)1522-726X(199905)47:13.0.CO;2-Z. PMID 10385166
- [Background] Gaspar J, Vonderwalde C, Hong MK, Eid-Lidt G, Almagor Y, Leon MB. [Stent coated with bovine pericardium: in vitro evaluation, in animals, and initial results in humans]. Arch Cardiol Mex. 2001 Oct-Dec;71(4):286-94. Spanish. PMID 11806031
- [Background] Gaspar J, Vonderwalde C, Eid-Lidt G. Treatment of coronary artery aneurysms by percutaneous sealing with bovine-pericardium-covered stents. Int J Cardiovasc Intervent. 1999;2(4):241-246. doi: 10.1080/acc.2.4.241.246. PMID 12623575
- [Result] Ferlini M, Russo F, Marinoni B, Repetto A, Canosi U, Ferrario M, Visconti LO, Bramucci E. Images in cardiology. Percutaneous coronary aneurysm obliteration using a novel pericardium-covered stent. J Am Coll Cardiol. 2010 Dec 14;56(25):2139. doi: 10.1016/j.jacc.2010.04.071. No abstract available. PMID 21144975